CLINICAL TRIAL: NCT06650878
Title: Randomized Controlled Trial Comparing the Desarda Tissue Technique With the Lichtenstein Technique in Primary Inguinal Hernia Repair
Brief Title: Desarda Tissue Technique vs Lichtenstein Technique for Primary Inguinal Hernia Repair
Acronym: HP-tis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Consorci Sanitari de l'Alt Penedès i Garraf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CSAPG-65
Record Dates: First submitted 2024-10-18; First posted 2024-10-21 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Inguinal Hernia Unilateral; Complications of Surgical Procedures or Medical Care
Keywords: Inguinal Hernia; lichtenstein technique; desarda technique
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Desarda Technique (Experimental): Patients asigned to this arm will be treated with Desarda Technique
  Interventions: Procedure: Desarda
- Lichtenstein Technique (Active Comparator): Patients asigned to this arm will be treated with Lichtenstein Technique
  Interventions: Procedure: Lichtenstein

INTERVENTIONS:
Procedure: Desarda — This technique prevent from using a mesh to surgical repair of a inguinal hernia
  Arms: Desarda Technique
Procedure: Lichtenstein — This technique implies using a mesh to surgical repair of a inguinal hernia
  Arms: Lichtenstein Technique

SUMMARY:
This study aims to evaluate whether a surgical technique (Desarda) is superior to the commonly used surgical technique (Lichtenstein) in inguinal hernia repair concerning the occurrence of postoperative complications. The Lichtenstein technique involves the use of a mesh, while the Desarda technique does not.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with primary inguinal hernia.
* Body mass index below 31
* Indication for inguinal hernia repair via anterior approach, either as outpatient surgery (CMA) or elective admission.
* Legal capacity to provide informed consent.

Exclusion Criteria:

* Patients with a weak, thin, or divided external oblique aponeurosis.
* Participants diagnosed with any of the following conditions:

  * Ongoing oncological disease
  * Cirrhotic patients classified as Child B or higher
* Women who have previously undergone a cesarean section
* Cognitive or affective conditions that limit the ability to cooperate with the study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 478 (Estimated)
Dates: Start 2025-03-26 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Rate of Participants with Post-surgery Complications | 3 months
  Any of the following complications: ● Sensation of a foreign body that persists beyond 3 months after surgery, self-reported by the participant ● Seroma within the first 30 days after surgery, verified through physical examination by a surgeon ● Hematoma within the first 30 days after surgery, verified through physical examination by a surgeon ● Infection at the surgical site within the first 30 days after surgery, verified by a surgeon ● Severe postoperative pain (7 or higher on the visual analog scale [VAS]) within the first 30 days after surgery, self-reported by the participant ● Chronic postoperative pain (persisting more than three months after surgery), self-reported by the participant ● Persistent loss of skin sensitivity beyond 30 days after surgery, self-reported by the participant ● Limitation of normal activities at home, outside the home, or at work beyond 3 months after surgery, self-reported by the participant

CONTACTS AND LOCATIONS:
Overall Officials: Javier Errando, MD, Principal Investigator — CSAPG
Locations (1):
- CSAPG, Sant Pere de Ribes, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
IPD (without personal identification data) could be shared by requirement from other researchers after the end of the study, and only for research purposes and previous approval of promotor center of the study (CSAPG). Anyway, Spanish and European Union legal policy about data protection will strictly be followed (IPD will not be transferred outside European Union).
Supporting Information: Study Protocol, ICF
Time Frame: After publication of main results of the study.
Access Criteria: IPD will be shared only for scientific research purposes and following the Spanish and European Union normative law about data protection. The requirements will be directed to the IP of the study. The IP will evaluate the request to verify and evaluate the data that is requested and the purposes for which it is requested. Next, the IP will transfer the request to the promotor center the study for the final decision.